CLINICAL TRIAL: NCT04896918
Title: Smoking, Snus Use and the Risk of COVID-19 in a Cohort of Adult Client of Public Dentistry Clinics: is There a Causal Association?
Brief Title: Tobacco Use and the Risk of COVID-19
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Norforsk (Unknown); Norwegian Institute of Public Health (Other Government); Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Maria Rosaria Galanti, Adjunct Professor, Karolinska Institutet
Other Study IDs: 4-1457/2021
Record Dates: First submitted 2021-05-20; First posted 2021-05-21 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Covid19
Keywords: Tobacco; Snus; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of adult client of public dental clinics in Region Stockholm: Tobacco use (cigarette smoking and/or snus use) will be considered as exposure. Information on tobacco use will be extracted by public dental clinic records in Stockholm Region (October 2015-January 2020). Any diagnosis of COVID-19, hospitalization, receiving intensive care, and death because of COVID-19 will be examined as outcomes. Diagnoses of COVID-19 will be obtained through record linkage with health care registers of inpatient and outpatient care (February 2020-August 2021).
  Interventions: Behavioral: Tobacco use

INTERVENTIONS:
Behavioral: Tobacco use

SUMMARY:
Contrasting hypotheses, including that of a protective role of nicotine, have been generated concerning the association between smoking and the occurrence of COVID-19 infection. The question has attracted a lively scientific and public debate. However, the studies conducted so far are based on clinical samples, with a majority of hospital case series, thus most likely suffering from bias due to selection.

The investigators propose to conduct an analysis of the potential causal association between smoking or the use of the Swedish smokeless tobacco snus and the occurrence of COVID-19 using data from a newly identified retrospective cohort in Sweden. Information on tobacco use will be extracted by public dental clinic records in Stockholm Region between October 2015 and January 2020. Information on diagnoses of COVID-19 will be obtained through record linkage with health care registers of inpatient and outpatient care during the period February 2020-August 2021. Socio-demographic information will be accrued from the register of the total population in Stockholm Region (Statistics Sweden). The risk of COVID-19 for tobacco users compared to non-tobacco users will be calculated as a measure of association adjusting for potential confounders.

DETAILED DESCRIPTION:
Background The role of tobacco use in the incidence and in the prognosis of the Severe acute respiratory syndrome-Cov2 disease (COVID-19 pandemic) has raised much international interest, due to contrasting findings reported so far in the scientific literature. On one side smoking may increase the risk of adverse outcomes in clinically overt COVID-19 requiring hospital admission. Several cross-sectional studies (case series) indicated a higher risk of negative disease progression among smokers compared to non-smokers in cases hospitalized with severe symptoms of the disease. On the other side, studies also suggest also that smoking is associated with a decreased risk of hospital admission with a diagnosis of COVID-19, or a decreased risk of occurrence of the disease in the community. These studies have noted 4 to 5 times lower proportions of smokers among patients hospitalized for COVID-19 compared with the underlying source population. A metanalysis of hospital case series confirmed this gap.

Given the public health importance of tobacco use as a risk factor for morbidity and mortality, it is urgent to provide both the scientific and the broad lay community with sound information from large population studies, something that the World Health Organization has also recommended.

Aim The present study aims to elucidate the potential causal association between tobacco use (smoking and snus) and COVID-19 using a population-based cohort study.

Methods In Sweden, the public dental clinics collect information at each visit on lifestyle and co-morbidities with relevance for oral health (health declaration), with a uniform instrument in use from October 2015. Smoking and snus use are ascertained as past use, current use and categories of intensity of current use. During February 2020 the usual routine activity of the clinics was disrupted by the pandemic, and the so-called oral health check-up was discontinued. About 450 000 adult clients of the public dentistry in Stockholm Region were identified in the period October 2015 to January 2020. Among these about 120000 were assessed within 7 months from the onset of the pandemic, therefore represent recent experiences. The investigators expect about 9% to be smokers and about 11% to be snus users. With the help of the national personal numbers assigned to every resident in Sweden at birth or at immigration, the investigators will link the reports of smoking among these clients with diagnoses of COVID-19 and other comorbidities registered in the regional database of inpatient and outpatient health care. The information in the dental clinic registers will be linked to the total population of the region of Stockholm, in order to extract socio-demographic information.

Statistical analysis plan The investigators will examine the role of tobacco use on the risk of the following events: any diagnosis of COVID-19, hospitalization, receiving intensive care, and death because of COVID-19 using generalized linear models, with and without possible confounders (age, gender, country of birth, type of employment, education and cohabitation), and within subgroups to identify potential effect modification (age group, gender [in analyses of snus use], assumed infection risk associated to occupation, pandemic period, and strategies of virologic testing, very restricted in the first 3 months, available on individual request thereafter).

ELIGIBILITY:
Inclusion Criteria:

* Being a client of the public dental clinics in the region of Stockholm (Sweden) between October 2015 and January 2020
* Being age 23 years or older
* Having tobacco use habits recorded in at least one visit

Exclusion Criteria:

* Not having a Swedish personal identity number
* Resident in assisted elderly dwelling

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult clients of the public dental clinics in Stockholm Region (Sweden) in the period between October 2015 and January 2020.
Sampling Method: Non-Probability Sample
Enrollment: 450000 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of COVID-19 | 18 months from the index case of the pandemic in Sweden
  Incident diagnoses of COVID-19, whether symptomatic or not, corresponding to a positive virologic test (PCR)
Hospital admission for COVID-19 | 18 months from the index case of the pandemic in Sweden
  Rates of hospital admission due to COVID-19 reported in the hospital register
Intensive unit care because of a diagnosis of COVID-19 | 18 months from the index case of the pandemic in Sweden
  Rates of admission to Intensive care units (IU) with a diagnosis of COVID-19 reported in the hospital register
Death for COVID-19 | 18 months from the index case of the pandemic in Sweden
  COVID-19 death rates where COVID-19 is mentioned as cause of death reported in the death register

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosaria Galanti, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Zhang JJ, Dong X, Cao YY, Yuan YD, Yang YB, Yan YQ, Akdis CA, Gao YD. Clinical characteristics of 140 patients infected with SARS-CoV-2 in Wuhan, China. Allergy. 2020 Jul;75(7):1730-1741. doi: 10.1111/all.14238. Epub 2020 Feb 27. PMID 32077115
- [Background] Dreher M, Kersten A, Bickenbach J, Balfanz P, Hartmann B, Cornelissen C, Daher A, Stohr R, Kleines M, Lemmen SW, Brokmann JC, Muller T, Muller-Wieland D, Marx G, Marx N. The Characteristics of 50 Hospitalized COVID-19 Patients With and Without ARDS. Dtsch Arztebl Int. 2020 Apr 17;117(16):271-278. doi: 10.3238/arztebl.2020.0271. PMID 32519944
- [Background] Rossato M, Russo L, Mazzocut S, Di Vincenzo A, Fioretto P, Vettor R. Current smoking is not associated with COVID-19. Eur Respir J. 2020 Jun 4;55(6):2001290. doi: 10.1183/13993003.01290-2020. Print 2020 Jun. PMID 32350106
- [Background] Farsalinos K, Barbouni A, Niaura R. Systematic review of the prevalence of current smoking among hospitalized COVID-19 patients in China: could nicotine be a therapeutic option? Intern Emerg Med. 2020 Aug;15(5):845-852. doi: 10.1007/s11739-020-02355-7. Epub 2020 May 9. PMID 32385628
- See also: Related Info — https://www.who.int/news-room/commentaries/detail/smoking-and-covid-19